CLINICAL TRIAL: NCT03148665
Title: A Prospective, Multi-site Trial of a Point of Care Saliva Based Detection Test Based on Soluble CD44 (OncAlert) for Presence of Disease in Previously Untreated Oral Cavity and Oropharynx Squamous Cell Carcinoma
Brief Title: Saliva-based Detection of CD44
Acronym: Detect 44
Status: Completed | Type: Observational
Sponsor: Joseph Califano (Other)
Collaborators: Vigilant Biosciences, Inc. (Industry); Greater Baltimore Medical Center (Other); San Diego Veterans Healthcare System (U.S. Federal Agency); NYU Langone Health (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor-Investigator, Joseph Califano, Study Chair, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: 161215
Record Dates: First submitted 2017-05-04; First posted 2017-05-11 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Oral Cavity Squamous Cell Carcinoma; Oropharynx Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Oropharynx; Squamous Cell Carcinoma of the Head and Neck
Keywords: Oral Cancer; Head and Neck Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Control population: Control population (n=150): absence of current or prior oropharyngeal carcinoma, no active cancer diagnosis. Control population includes at least 50 subjects who have smoked at least 100 cigarettes during lifetime OncAlert saliva-based screening, a noninvasive point of care salivary rinse test performed as a one-time test for control subjects
  Interventions: Device: OncAlert
- Cancer population: Cancer population (n=150): patients with previously untreated oral cavity or oropharynx squamous cell carcinoma with absence of distant metastasis OncAlert saliva-based screening, a noninvasive point of care salivary rinse test performed as at pretreatment and post treatment 3,6, 12, and 18 month time points in oral cavity/oropharynx cancer patients
  Interventions: Device: OncAlert

INTERVENTIONS:
Device: OncAlert — A noninvasive point of care salivary rinse test performed as 1) a one-time test for control subjects, 2) at pretreatment and post treatment 3,6, 12, and 18 month time points in oral cavity/oropharynx cancer patients

SUMMARY:
The purpose of this study is to test the ability of OncAlert™ to screen for cancer and the reappearance of cancer. OncAlert™ was developed by Vigilant Biosciences, a collaborator in this research study. OncAlert™ is an oral rinse which is spit into a cup and sent to a laboratory for analysis. OncAlert™ is considered experimental by the FDA because it is not approved for the screening of cancer.

DETAILED DESCRIPTION:
A noninvasive point of care salivary rinse test performed as 1) a one-time test for control subjects, 2) at pretreatment and post treatment 3,6, 12, and 18 month time points in oral cavity/oropharynx cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Patient has the ability to understand and the willingness to sign a written informed consent.
* Previously untreated, measurable squamous cell carcinoma of the oral cavity or oropharynx with no evidence of distant metastasis, T1-4N0-3M0
* No prior history of treated upper aerodigestive tract cancer
* No concurrent, second, active malignancy other than oral cavity and/or oropharynx cancer
* Planned to undergo treatment with curative intent
* Able to follow up after therapy at 3, 6, 12, and 18 months after completion of therapy during routine post treatment follow up
* For control subjects: no evidence or history of upper aerodigestive tract cancer
* For control subjects: absence of any suspected or confirmed active malignancy at time of enrollment
* Patients may have had prior therapy for malignancy other than upper aerodigestive malignancy completed 2 years prior to enrollment if they have been disease free since completion of therapy
* Patient is ≥ 18 years of age.
* Both men and women of all races and ethnic groups are eligible for this trial.
* Performance Status ≤ ECOG 3
* Patient is able to gargle and spit 5 cc of saline
* Patients may be concurrently enrolled in other therapeutic or detection clinical trials

Exclusion Criteria:

* Prior completed therapy for an upper aerodigestive tract cancer within the past 3 years.
* Patient unable to gargle and spit 5 cc of saline, or anticipated to be unable to gargle and spit after completion of therapy
* Patient unable or does not intend to undergo curative therapy
* Patient with concurrent, second primary malignancy under active therapy or completed therapy within 2 years prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer patients were identified through tumor board. Control patients were identified by referral.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
To validate performance of the Vigilant Oral Rinse Point of Care strip in a multi-institutional clinical setting | 4 years
  * The agreement between CD44 ELISA and BCA test as measured using the POC test (OncAlert) and central laboratory testing at Vigilant The concordance of these two measures will be assessed using Cohen's kappa statistic for a dichotomized outcome (positive vs. negative test). A kappa of 0.6 or lower will be considered of insufficient concordance, and the minimum required level indicating adequate concordance is a kappa of 0.8
  * The sensitivity and specificity of the OncAlert test to detect OOPSCC in cases compared to a non cancer control population.
  * A specificity of 0.65 minimally acceptable for the Vigilant POC test. In order to demonstrate a clinically acceptable level of specificity, a performance goal of 0.75 is chosen

SECONDARY OUTCOMES:
To prospectively validate the performance of pretreatment Vigilant Oral Rinse Point of Care strip and Sol CD44 as a predictor of outcome for oral/oropharyngeal cancer in a point of care multi-institutional clinical setting | 4 years
  - The association of salivary CD44 POC test biomarkers, including both the POC test and quantitative ELISA based assay with clinical characteristics of OOPSCC patients, such as site, stage, treatment, smoking, alcohol, HPV status, and patient overall and disease free survival using univariate and multivariate analyses.
To determine the association of post treatment salivary solCD44 and the Vigilant Oral Rinse Point of Care strip with disease outcome in oral/oropharyngeal cancer | 4 years
  - The association of salivary CD44 POC test biomarkers, including both the POC test and quantitative ELISA based assay with recurrence of OSCC in an OSCC population with clinical characteristics of OOPSCC patients, such as site, stage, treatment, smoking, alcohol, HPV status, and patient overall and disease free survival using univariate and multivariate analyses and determine the magnitude of that association.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Califano, MD, Study Chair — University of California, San Diego
Locations (4):
- United States (4):
  - UCSD Moores Cancer Center, La Jolla, California
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - New York University College of Dentistry, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franzmann EJ, Qi Y, Peifer S, Messer K, Messing B, Blanco RG, Khan Z, Fahkry C, Coffey C, Califano J 3rd. Salivary CD44 and Total Protein Levels to Detect Risk for Oral and Oropharyngeal Cancer Recurrence: A Nonrandomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Oct 1;150(10):843-850. doi: 10.1001/jamaoto.2024.2490. PMID 39145961